CLINICAL TRIAL: NCT02287337
Title: Validation of a Clinical Prediction Rule to Identify Patients With Neck Pain Likely to Benefit From Cervical Spine Manipulation: A Randomized Clinical Trial
Brief Title: Validation of CPR for Manipulation for Neck Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB approval expired when PI left UNLV
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Emilio J Puentedura, PT, DPT, PhD, Associate Professor, University of Nevada, Las Vegas
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UNLV-1212-4327
Record Dates: First submitted 2014-11-03; First posted 2014-11-10 (Estimated); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Cervicalgia
Keywords: Neck pain
MeSH Terms: conditions — Neck Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manipulation (Experimental): Patients will receive cervical manipulation on 2 visits and then a further 3 visits of therapeutic exercises
  Interventions: Procedure: Manipulation; Procedure: Exercise
- Exercise (Other): Patients will receive 5 visits of therapeutic exercises
  Interventions: Procedure: Exercise

INTERVENTIONS:
Procedure: Manipulation — High velocity low amplitude thrust joint manipulation to cervical spine facet joints
  Arms: Manipulation
Procedure: Exercise — Therapeutic exercises to the cervical, thoracic and scapular musculature

SUMMARY:
The purpose of this study is to see if a recently developed clinical prediction rule (CPR) will successfully identify which patients with neck pain will respond rapidly and favorably to manipulation of their cervical spine.

DETAILED DESCRIPTION:
Consenting patients with a primary complaint of neck pain will be screened for contraindications to cervical spine manipulation and if eligible to participate in the study, will undergo a detailed subjective (history) and objective (physical) examination. At the completion of the examination, they will be assigned to one of two treatment arms - cervical manipulation and exercise or exercise only. They will receive up to 5 treatment sessions and be followed at 1 month, 3 months and 6 months after initial visit.

ELIGIBILITY:
Inclusion Criteria:

* Primary complaint of mechanical neck pain with or without unilateral upper extremity symptoms (mechanical neck pain is defined as neck pain/ symptoms that are altered/ affected by activity, movement and posture)
* NDI score at least 10 points out of 50.

Exclusion Criteria:

* Red flags noted in the patient's Neck Medical Screening Questionnaire (i.e. tumor, fracture, metabolic diseases, Rheumatoid Arthritis, osteoporosis, prolonged history of steroid use, etc.)
* History of whiplash injury within the past six weeks
* Diagnosis of cervical spinal stenosis or bilateral upper extremity symptoms
* Evidence of central nervous system involvement, to include hyperreflexia, sensory disturbances in the hand, intrinsic muscle wasting of the hands, unsteadiness during walking, nystagmus, loss of visual acuity, impaired sensation of the face, altered taste, the presence of pathological reflexes (i.e. positive Hoffman's and/or Babinski reflexes), etc.
* Two or more positive neurologic signs consistent with nerve root compression, including any two of the following: a. Muscle weakness involving a major muscle group of the upper extremity b. Diminished upper extremity muscle stretch reflex (biceps brachii, Brachioradialis, or triceps reflex) c. Diminished or absent sensation to pinprick in any upper extremity dermatome
* Prior surgery to the neck or thoracic spine
* Pending legal action regarding their neck pain
* Insufficient English language skills to complete all questionnaires
* Inability to comply with treatment and follow-up schedule

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2017-08-26 (Actual); Study Completion 2017-08-26 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index | 6 months
  10-item patient self-report measure of perceived disability

SECONDARY OUTCOMES:
Medication Use | 6 months
Global Rating of Change Scale | 6 months
Numeric Pain Rating Scale | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nevada Las Vegas, Las Vegas, Nevada, United States